CLINICAL TRIAL: NCT04357535
Title: Prognosis of SARS-Cov 2 Positive Patients Receiving Angiotensin Converting Enzyme Inhibitors (ACE-I) and Angiotensin II Receptor Antagonists (ARBs)
Brief Title: Prognosis of Coronavirus Disease 2019 (COVID-19) Patients Receiving Receiving Antihypertensives
Status: Completed | Type: Observational
Sponsor: Hakeam Abdulaziz Hakeam (Other)
Collaborators: Buraidah Central Hospital (Other Government); King Khalid University Hospital (Other); Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Sponsor-Investigator, Hakeam Abdulaziz Hakeam, Clinical Pharmacy Specialist, Surgery. Pharmaceutical Care Division, King Faisal Specialist Hospital & Research Centre. Adjunct Assistant Clinical Professor College of Medicine, Alfaisal University., King Faisal Specialist Hospital & Research Center
Organization: King Faisal Specialist Hospital & Research Center (Other)
Other Study IDs: 2210061
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: Coronavirus Disease 2019; Angiotensin Converting Enzyme Inhibitors; Angiotensin II Receptor Blockers
MeSH Terms: conditions — COVID-19 | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Primary Cohort: Patients enrolled in this study will have data collected from the beginning of their hospital stay until discharge.
  Data collected will include:
  * Patient demographics (age, sex, weight, and height)
  * Indication for ACE-I, ARB therapy, duration and doses
  * Use of any a non ACE-I/ ARB sntihypertensive agents
  * Comorbidities, and COVID19 related markers: Including WBC, plateltes, ferritin, CRP, CK, and LD
  * CT scan reports
  * First positive COVID19 PCR
  * Admission to the intensive care unit (ICU) and data relating to ICU stay.
  Interventions: Drug: Angiotensin-Converting Enzyme Inhibitors (ACE-I) and Angiotensin II Receptor Blockers (ARB)

INTERVENTIONS:
Drug: Angiotensin-Converting Enzyme Inhibitors (ACE-I) and Angiotensin II Receptor Blockers (ARB) — ACE-I and ARB are a class of blood pressure lowering medications used to manage hypertension.
  Other Names: ACE-I; ARB

SUMMARY:
Coronavirus disease 2019 (COVID-19) ,caused by the newly identified Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) virus, has shown substantial global spread affecting over 2 million people and claiming over 120,000 lives to date. In March 2020, the World Health Organization (WHO) declared COVID-19 a global pandemic. The spectrum of manifestations of COVID19 infection ranges from mild flu-like symptoms to severe acute respiratory distress syndrome (ARDS), with an associated fatality rate of 1.4%. The suggested mode of entry of the SARS-CoV-2 into the human respiratory epithelium is through the angiotensin-converting enzyme 2 (ACE2) protein expressed on alveolar cell surfaces. This entry mechanism has sparked the interest of the scientific community. Preliminary epidemiological reports showed an increased risk of ARDS in hypertensive COVID-19 patients. This leads to the hypothesis that hypertensives treated with angiotensin-converting enzyme inhibitor (ACE-I) are at an increased risk of developing complicated COVID-19 infections . Other studies have refuted these claims as unsupported. Studies revealing the up regulation of ACE2 in cells of patients treated with ACE-I or ARBs were the underlying foundation for these claims. This study aims to assess the impact of ACE-I and/or ARBs on the prognosis of patients with COVID19.

DETAILED DESCRIPTION:
Design and Patients: this is a prospective, observational multi-center study, to be conducted at King Faisal Specialist Hospital and Research Centre (KFSH & RC), Riyadh, Saudi Arabia as a primary center. Collaborating centers are Buraidah Central hospital,King Khalid University Hospital and King Abdullah bin Abdulaziz University Hospital (affiliate of Princess Nourah Bint Abdulrahman University)

Sample size: 226 subjects.

Protocol: Patients diagnosed with COVID19 infection via positive polymerase chain reaction (PCR) test will be screened for one of the following five comorbidity (hypertension, diabetes mellitus, cerebrovascular disease, coronary artery disease, and heart failure) will be identied on admission to hospital. The use of ACE-I and ARBs or other antihypertensive medications will be recorded. Additional information to be gathered will include the following: patient demographics (age, sex, weight, and height), indication for ACE-I or ARB therapy, duration therapy and doses; plasma or serum levels of the following laboratories will be obtained on admission: creatinine levels, lactate dehydrogenase, creatinine kinase, ferritin, D-Dimer, and c-reactive protein. The date of positive COVID19 PCR; admission to the intensive care unit (ICU) with calculating the Sequential Organ Failure Assessment (SOFA) score. The requirement of mechanical ventilation and vasopressors will be recorded with a length of ICU stay. Patients fulfilling the criteria of acute respiratory distress (ARDS) will be recorded, and the PF ratio will be assessed for all subjects admitted to the ICU. Patient who die in ICU or during hospitalization will be recorded. The entirety of the hospitalization period will be determined and recorded.

Outcome Assessment: The primary endpoint will be the severity of COVID-19 infection, described as the composite of admission to the intensive care unit, requirement for invasive mechanical ventilation or death. The use of ACE-I and ARBs will be assessed independently for associations with severity of respiratory disease.

The rate of patients using ACE-I or ARBs will be reported with the indications for their use. The association of ACE-I or ARBs with prognosis of patients with COVID19 will be reported.

ELIGIBILITY:
Inclusion Criteria:

Criteria Include patients infected with the COVID19 (via positive PCR) aged ≥ 18 years with one of the following:

* Hypertension
* Coronary artery disease
* Heart failure
* Diabetes mellitus.

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include patients admitted in King Faisal Specialist Hospital and Reseach Centre (KFSH&RC) Riyadh, Saudi Arabia.
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Severity of COVID-19 Infection | From date of study enrolment until discharge from hospital or death from any cause, whichever came first, assessed up to 4 weeks.
  Admission to intensive care unit, requirement for invasive ventilation or death

SECONDARY OUTCOMES:
Degree of severity of respiratory disease | From date of study enrolment until discharge from hospital or death from any cause, whichever came first, assessed up to 4 weeks.
  PaO2/FiO2 ratio (PF) ratio
Septic shock as defined by sepsis-3 criteria | From date of study enrolment until discharge from hospital or death from any cause, whichever came first, assessed up to 4 weeks.
  Defined as sepsis with hypotension requiring vasopressors to maintain mean arterial pressure (MAP) 65 mm Hg and having a serum lactate level >2 mmol/L (18 mg/dL) despite adequate volume resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Hakeam A Hakeam, MSPharm BCPS, Principal Investigator — King Faisal Specialist Hospital and Research Centre (KFSH&RC)
Locations (1):
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
On publication, according to the journal requirements

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Patel AB, Verma A. COVID-19 and Angiotensin-Converting Enzyme Inhibitors and Angiotensin Receptor Blockers: What Is the Evidence? JAMA. 2020 May 12;323(18):1769-1770. doi: 10.1001/jama.2020.4812. No abstract available. PMID 32208485
- [Background] Esler M, Esler D. Can angiotensin receptor-blocking drugs perhaps be harmful in the COVID-19 pandemic? J Hypertens. 2020 May;38(5):781-782. doi: 10.1097/HJH.0000000000002450. No abstract available. PMID 32195824
- [Derived] Hakeam HA, Alsemari M, Duhailib ZA, Ghonem L, Alharbi SA, Almutairy E, Sheraim NMB, Alsalhi M, Alhijji A, AlQahtani S, Khalid M, Barry M. Association of Angiotensin-Converting Enzyme Inhibitors and Angiotensin II Blockers With Severity of COVID-19: A Multicenter, Prospective Study. J Cardiovasc Pharmacol Ther. 2021 May;26(3):244-252. doi: 10.1177/1074248420976279. Epub 2020 Nov 24. PMID 33231487
- See also: World Health Organization Data — http://www.who.int/emergencies/diseases/novel-coronavirus-2019